CLINICAL TRIAL: NCT03100032
Title: A Prospective Multi-centre, Randomised, Controlled Study to Evaluate the Safety and Preliminary Effectiveness of NVD-001 for the Treatment of Low Grade Degenerative Lumbar Spondylolisthesis by Interbody Fusion (L1 - S1)
Brief Title: Safety and Preliminary Effectiveness of NVD-001 for the Treatment of Low Grade Degenerative Lumbar Spondylolisthesis
Acronym: Spine1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novadip Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NVD-CLN01; 2016-002642-23 (EudraCT Number)
Record Dates: First submitted 2017-02-08; First posted 2017-04-04 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-06

CONDITIONS: Spondylolisthesis
Keywords: Spinal Fusion; Lumbar Interbody Fusion; Autologous Stem Cell Therapy; Bone Graft; Demineralized Bone Matrix; Polyetheretherketone (PEEK) cage
MeSH Terms: conditions — Spondylolisthesis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVD-001 (Experimental): Autologous osteogenic cells in ECM with DBM
  Interventions: Biological: NVD-001
- Standard of Care (Active Comparator): Best standard of care in surgical practice
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Biological: NVD-001 — At the Investigator's discretion, one or two interbody polyetheretherketone (PEEK) cage(s) filled and surrounded with NVD-001.
  Arms: NVD-001
Procedure: Standard of Care — At the Investigator's discretion, one or two interbody polyetheretherketone (PEEK) cage(s) filled and surrounded with autologous locally cancellous bone (laminectomy)
  Arms: Standard of Care

SUMMARY:
A prospective multi-centre, randomised, controlled study to evaluate the safety and preliminary effectiveness of NVD-001 for the treatment of low grade degenerative lumbar spondylolisthesis by interbody fusion (L1 - S1).

DETAILED DESCRIPTION:
This is a prospective multi-centre, randomised, controlled study to evaluate the safety and preliminary effectiveness of NVD-001 for the treatment of low grade degenerative lumbar spondylolisthesis by interbody fusion of one vertebral segment (L1-S1). The study consists of a 12-month initialfollow-up period post-surgery and a subsequent 12-month long term follow-up.

NVD-001 is an autologous cellular medicinal product obtained by culture of adipose tissue (liposuction) leading to osteogenic cells after ex vivo isolation, expansion and differentiation of pluripotent adipose-tissue stem cells (ASC), and combination with an allogeneic fully demineralised bone matrix into a 3D bone implant.

Patients diagnosed with symptomatic degenerative spondylolisthesis grade I or II with an indication for spinal fusion of one vertebral segment (L1-S1) who sign informed consent and are eligible will be randomised either to the experimental group (surgical intervention for spinal lumbar interbody fusion with NVD-001) or to the control group (commonly used surgical intervention for spinal lumbar interbody fusion (TLIF, PLIF, minimally invasive or open approach) with one or two PEEK cage(s) filled and surrounded by locally harvested autologous cancellous bone (laminectomy).

ELIGIBILITY:
Inclusion Criteria:

Any subject meeting all of the following inclusion criteria and verified by the Investigator during the screening period:

* Subject has understood and accepted to participate in the study according to all study procedures by signing the approved informed consent.
* Male or female subjects aged >18 and is skeletally mature (epiphyses closed).
* Subject has clinically important pain or neurological symptoms with or without claudication due to symptomatic degenerative spondylolisthesis grade I or II (Meyerding Classification).
* Conservative treatment of disease has failed for at least 3 months since diagnosis. (ISASS 2011)
* Subject has a preoperative ODI score >30.
* Subject has an indication for spinal fusion of one vertebral segment (L1-S1) due to symptomatic degenerative spondylolisthesis grade I or II diagnosed by computed tomography (CT) scan and/or magnetic resonance imaging (MRI) and/or dynamic radiography.
* Subject is suitable for surgical operation and incorporation of the PEEK cage(s) by transforaminal lumbar interbody fusion (TLIF) or posterior lumbar intervertebral fusion (PLIF) by minimally invasive or open approach in one mobile segment (L1- S1) with bilateral rigid fixation. No posterolateral lumbar fusion (PLF) technique is allowed.
* Subject is, in the Investigator's opinion, psychosocially, mentally and physically able to fully comply with this protocol, including the postoperative regimen and follow-up visits.
* At screening, local laboratory safety test results are clinically acceptable and serology results for HIV, HBV, HCV, HTLV I/II and syphilis are in accordance with country specific requirements for donation of Human Body Material. At time of adipose tissue collection, central laboratory serology and molecular test panel for HIV, HBV, HCV, HTLV I/II and syphilis must be in accordance with Belgian specific requirements for release of Human Body Material.
* Women of childbearing potential (WOCBP) including peri-menopausal women who have had a menstrual period within 1 year prior to surgery have to have a negative pregnancy test. Results have to be available and negative for the patient to be entered in the study.
* WOCBP have to use an effective method of birth control 2 months prior to study entry or to surgical intervention date and throughout the study duration (defined as a method which results in a failure rate of less than 1% per year) such as:

  * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomised partner (provided that partner is the sole sexual partner of the trial participant and that the surgical success of vasectomy has been confirmed)
  * Sexual abstinence For each case of delayed menstrual period, confirmation of absence of pregnancy is strongly recommended. This recommendation also applies to WOCBP with infrequent or irregular menstrual cycles. In case a urine pregnancy test is positive, a confirmatory blood pregnancy test is obligatory.

Exclusion Criteria:

Any subject meeting any of the following exclusion criteria verified by the Investigator during the screening period will be excluded from enrolment into the study.

* Subject has known history of hypersensitivity or anaphylactic reaction to PEEK.
* Due to medical or other reasons spine fusion cannot be delayed for up to 6 months.
* Indications for spinal fusion other than symptomatic degenerative spondylolisthesis grade I and II (Meyerding Classification).
* Subject displays drug or alcohol dependence, serious current illness, mental illness or extenuating circumstance or any other factors which, in the opinion of the Investigator, will interfere with study conduct or interpretation of the results.
* Subject has documented metabolic disease such as but not limited to severe osteoporosis, osteogenesis imperfect, or osteomalacia.
* Subject with poorly controlled diabetes mellitus as assessed by glycohaemoglobin (HbA1c) > 8% (at least 2 values per year for last 2 years)
* Subject is underweight, i.e. body mass index (BMI) ≤18.5 or has a BMI of ≥40, or ≥35 and experiencing obesity-related health conditions, such as high blood pressure or diabetes at V0a.
* Overt or active local or systemic infection, including latent infection around (area of) the future surgical implant site.
* Subject has a history of previously attempted spinal fusion at the same level, or spine level immediately adjacent to the level to be operated on in this study. Decompressive surgery alone (laminectomy) is not an exclusion criterion.
* Subject is on a transplant list or having received a solid organ transplant at any point in the past.
* Pregnant or breast-feeding woman.
* Involved in or planning to engage in litigation related health problems.
* Subject is a prisoner.
* Subject had an acute fracture of the spine within 6 months prior V0a in the study.
* Subject is known to require additional surgery to the lumbar spinal region within the next 2 years after enrolment in the study.
* Subject is currently taking chronically any medications that might affect bone metabolism or the quality of bone formation such as but not limited to bisphosphonates, steroids, methotrexate, anticoagulant therapies, immunosuppressants or immunotherapy.
* Subject is currently using an electrical bone growth stimulator
* Subject is positive for human immunodeficiency virus (HIV) 1 or 2, hepatitis B (HBsAg or PCR positive) or C, human T-cell lymphotropic virus (HTLV) 1 or 2, or syphilis at screening (V0a).
* Subject was exposed to any experimental therapy with another investigational drug within 60 days prior to screening or enrolment in any concurrent study that may confound the results of this study.
* Subject previously received a cellular therapy (at any point in time).
* Subject was exposed to therapy for a malignancy or pre-malignant entity, and not confirmed disease-free for 5 years or more.
* Any clinically relevant chronic disease associated with renal or hepatic insufficiency or any chronic disease of such severity that surgery could be detrimental to the survival of the patient.
* Any other illness which might reduce life expectancy to less than 2 years from screening.
* Subject is on chronic immunosuppressive therapy (immunosuppressants/immunotherapy) due to inflammatory or systemic disease.
* Subject has an active inflammatory systemic autoimmune disease that could interfere with bone metabolism such as but not limited to rheumatoid arthritis, ankylosing spondylarthritis, inflammatory bowel disease, systemic lupus erythematosus or thyroid diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01; Primary Completion 2021-01 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
NVD-001 (nocc AEs) | 12 months
  Number of Adverse Events (AEs) severity, relatedness to the product or procedure, required action and outcome, up to 12 months post-surgery
NVD-001 (npat AEs) | 12 months
  Number of participants presenting Adverse Events (AEs).
NVD-001 (nocc SAEs) | 24 months
  Number of serious Adverse Events (SAEs), severity, relatedness to the product or procedure, required action and outcome.
NVD-001 (npatSAEs) | 24 months
  Number of participants presenting Serious Adverse Events (AEs).
NVD-001 (nocc AESI) | 24 months
  Number of Adverse Events of Special Interest (AESI) using lumbar spine CT and radiographic images.
NVD-001 (npat AESI) | 24 months
  Number of participants with Adverse Events of Special Interest (AESI) using lumbar spine CT and radiographic images.
NVD-001 (npat Safety X-rays) | 24 months
  Number of participants with appearance or absence of calcification/ ossification and ectopic bone formation in comparison with preoperative, as determined by chest X-rays.
NVD-001 (npat Safety Post-Op) | 1 month
  Number of participants with occurrence or absence of surgical intervention-related safety parameters such as infection and peri- and post-operative blood loss volume

SECONDARY OUTCOMES:
NVD-001 (LSF) | 24 months
  Lumbar Spine Fusion progression and non-fusion assessed by serial CT-Scans images of lumbar spine post-surgery and lumbar spine static and dynamic radiographic images.
NVD-001 (ODI) | 24 months
  Functional disability by means of Oswestry Disability Index (ODI).
NVD-001 (BPI) | 24 months
  Pain by means of Brief Pain Inventory (BPI).
NVD-001 (OTE) | 24 months
  Overall treatment effect using OTE scale.
NVD-001 (QoL) | 24 months
  Quality of life (QoL) by means of patient's questionnaire EuroQoL 5 Dimensions post-surgery.
NVD-001 (timeSurgery) | 1 day
  Surgical duration.
NVD-001 (stayPostOp) | 7 days
  Duration of postoperative hospital stay.
NVD-001 (subsequentSurgery) | 24 months
  Description of subsequent surgical interventions (revision, removal, reoperation and supplemental fixation).

CONTACTS AND LOCATIONS:
Overall Officials: Denis Dufrane, MD, PhD, Study Director — Novadip Biosciences; Christian Raftopoulos, MD, PhD, Principal Investigator — Saint-Luc University Hospital, Department of Neurosurgery
Locations (12):
- Belgium (6):
  - Hôpital Erasme - Neurosurgery Department, Brussels
  - Universitair ziekenhuis Brussel - Brussels Health Campus - Department of Orthopaedics and Traumatology, Brussels
  - Saint-Luc University Hospital, Brussels
  - Algemeen Ziekenhuis Monica O.L.V. - Campus Deurne, Deurne
  - Ziekenhuis Oost-Limburg, Campus Sint-Jan, Genk
  - Centre Hosp. Univ. UCL - Namur site Godinne - Service de neurochirurgie, Yvoir
- Czechia (2):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice v Motole, Prague
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne Angelius Provita, Katowice
  - Szpital Św. Rafała, Krakow
  - Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im. W. Degi Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion, coded data, in European Clinical Trial registry (https://www.clinicaltrialsregister.eu)